CLINICAL TRIAL: NCT01635595
Title: AdCa of the Esophagus and Cardia (ADEC): Relationship Between Nodal Metastasization and the Presence Absence of Intestinal Metaplasia in the Esophagus and Stomach
Brief Title: Nodal Status in Adenocarcinoma of the Esophagus an Cardia
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor, University of Bologna
Other Study IDs: Cardia AdCa UNIBO
Record Dates: First submitted 2012-07-03; First posted 2012-07-09 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastric Cardia
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Esophagectomy; Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with BIM: Patients affected by adenocarcinoma of the distal esophagus and cardia with preoperative diagnosis of BIM underwent subtotal esophagectomy and gastric pull up.
  Interventions: Procedure: Subtotal esophagectomy and gastric pull up
- Patients without BIM: Patients affected by adenocarcinoma of the distal esophagus and cardia without preoperative diagnosis of BIM underwent subtotal esophagectomy at the azygos vein, total gastrectomy and esophagojejunostomy.
  Interventions: Procedure: Subtotal esophagectomy at the azygos vein, total gastrectomy

INTERVENTIONS:
Procedure: Subtotal esophagectomy and gastric pull up — Subtotal esophagectomy and gastric pull up and radical thoracic (2,3,4R,7,8,9)and abdominal (15,16,17,18,19,20) lymphadenectomy
  Other Names: Esophagectomy
  Groups: Patients with BIM
Procedure: Subtotal esophagectomy at the azygos vein, total gastrectomy — Subtotal esophagectomy at the azygos vein, total gastrectomy and esophagojejunostomy and radical thoracic (2,3,4R,7,8,9) abdominal (15,16,17,18,19,20) lymphadenectomy.
  Other Names: Esophagectomy; Gastrectomy
  Groups: Patients without BIM

SUMMARY:
Adenocarcinoma of the distal esophagus and cardia are grouped among the thoracic tumors according to the TNM 7th ed., however controversy is pending on the unique or dual pathogenesis (GERD or gastric-like cancerogenesis). It has been shown that biological patterns differ according to the presence (+) or absence (-) of Barrett's epithelium (BIM) and gastric intestinal metaplasia (GIM) in the fundus and antrum. Lymphatic metastatic spreading may differ according to the type of tumor. The investigators retrospectively investigated the pathways of lymphatic spreading in 194 consecutive patients who received radical surgery for adenocarcinoma of the esophagus and cardia with or without BIM and GIM.

DETAILED DESCRIPTION:
The assumption that adenocarcinoma of the esophagus and cardia (ADEC) originates only from the sequence intestinal metaplasia followed by dysplasia and cancer is controversial. It has been shown that biological patterns differ according to the presence (+) absence (-) of Barrett's epithelium (BIM) and of gastric intestinal metaplasia (GIM) in the fundus and antrum. Lymphatic metastatic spreading may differ according to the type of tumor.

Preoperatively patients underwent histological search for Barrett's esophagus (BIM) in mucosa surrounding (ADEC) and intestinal metaplasia in the gastric corpus and antrum mucosa (GIM). Patients in which BIM was documented underwent sub total esophagectomy and gastric pull up (group 1), others underwent esophagectomy at the azygos vein + total gastrectomy with Roux Y esophagojejunostomy (group 2). Radical lymphadenectomy was identical in both procedures except for the greater curvature station.

ELIGIBILITY:
Inclusion Criteria:

* preoperative diagnosis of adenocarcinoma of the distal esophagus and cardia
* preoperative from local to locally advanced disease
* absence of neoadjuvant therapy

Exclusion Criteria:

* neoadjuvant therapy
* metastatic disease
* unfit for surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a preoperative diagnosis of adenocarcinoma of the distal esophagus and cardia who underwent surgery up to December 2011, which fully adhered to the pre and postoperative protocol, including endoscopic gastric mucosa sampling.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2006-01; Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Mattioli, Prof., Principal Investigator — University of Bologna
Locations (1):
- Division of Thoracic Surgery, Center for the Study and Therapy of Diseases of the Esophagus. Alma Mater Studiorum - University of Bologna, GVM Care & Research, Maria Cecilia Hospital, Cotignola, Ravenna, Italy

REFERENCES:
- [Background] Mattioli S, Di Simone MP, Ferruzzi L, D'Ovidio F, Pilotti V, Carella R, D'Errico A, Grigioni WF. Surgical therapy for adenocarcinoma of the cardia: modalities of recurrence and extension of resection. Dis Esophagus. 2001;14(2):104-9. doi: 10.1046/j.1442-2050.2001.00165.x. PMID 11553218
- [Result] Mattioli S, Ruffato A, Di Simone MP, Corti B, D'Errico A, Lugaresi ML, Mattioli B, D'Ovidio F. Immunopathological patterns of the stomach in adenocarcinoma of the esophagus, cardia, and gastric antrum: gastric profiles in Siewert type I and II tumors. Ann Thorac Surg. 2007 May;83(5):1814-9. doi: 10.1016/j.athoracsur.2007.01.016. PMID 17462405